CLINICAL TRIAL: NCT06542133
Title: AVEIR Remote Care System Data Collection Non-Significant Risk Study
Brief Title: AVEIR Remote Care System Non-Significant Risk Study
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10527
Record Dates: First submitted 2024-07-18; First posted 2024-08-07 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Pacemaker; Cardiac Rhythm Disorder; Bradycardia
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Observational, Single Arm, Non Randomized: Aveir leadless pacemaker system patients
  Interventions: Device: AVEIR remote care system

INTERVENTIONS:
Device: AVEIR remote care system — In-clinic or an at-home system designed to support remote follow up in Aveir leadless pacemaker patients

SUMMARY:
The goal of the study is to understand the performance of the AVEIR Remote Care System in an initial patient cohort which will inform the ability to offer a remote follow-up solution to all patients implanted with Aveir LP devices.

DETAILED DESCRIPTION:
To collect acute performance data about the AVEIR Remote Care System in participants implanted with a compatible dual or single chamber Aveir Leadless Pacemaker System by participants completing remote transmissions with the system

ELIGIBILITY:
Inclusion Criteria:

* Subject must provide written informed consent prior to any study-related procedure.
* Subject is willing and has consented to study clinical procedure.
* Subject is ≥ 18 years of age or age of legal consent, whichever age is greater
* Subject has an active, appropriately functioning Aveir leadless pacemaker system
* Subject is willing to use the device

Exclusion Criteria:

* Subject is unable to read/write at a sufficient level to provide informed consent.
* Subject is unable to make the decision to participate in a clinical investigation on their own or are unable to fully understand all aspects of the investigation that are relevant to the decision to participate.
* Subject has presence of medical, social, or psychological conditions that, in the investigator's opinion, could confound the study, limit the subject's ability to participate in the clinical investigation .

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Successful end-to-end transmission performance metrics | The expected duration of each subject's participation is approximately 30 minutes for an in-clinic visit to complete two transmissions and thereafter an optional at-home transmission (expected duration 10-15 minutes)
  Successful transmission performance metrics of the AVEIR Remote Care System in approximately 32 subjects who have received an Aveir LP implanted system as part of their standard of care.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Premier Cardiology, Inc, Newport Beach, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sundaram S, Chellappa N, Chaniary K, Lo M, Nair D, Banker R. Remote monitoring of leadless pacemakers using a novel conductive telemetry communication method. J Interv Card Electrophysiol. 2025 Jul 22. doi: 10.1007/s10840-025-02095-8. Online ahead of print. PMID 40694240